CLINICAL TRIAL: NCT01135082
Title: The Immunogenicity and Safety of Pneumococcal Conjugate Vaccine in Human Immunodeficiency Virus - Infected Children
Brief Title: Pneumococcal Conjugate Vaccine (PCV) in HIV- Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Pediatric infectious diseases section, King Chulalongkorn Memorial hospital, Chulalongkorn University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 135
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: HIV
Keywords: immunogenicity; safety; Pneumococcal conjugate vaccine; HIV infected children; objective of this study is to assess the safety and immunogenicity of a 7 - valent PCV vaccine among HIV - infected compared with HIV - exposed children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Receive valent pneumococcal conjugated vaccine in HIV - infected children
  Interventions: Biological: valent pneumococcal conjugated vaccine
- 2 (Other): Receive valent pneumococcal conjugated vaccine in HIV negative children
  Interventions: Biological: valent pneumococcal conjugated vaccine

INTERVENTIONS:
Biological: valent pneumococcal conjugated vaccine — Dosage: 0.5 ml per dose Administration: intramuscular injection Location: left deltoid area x 1 injection Frequency: depend on first dose of vaccination. If 2-6 months of age, vaccination at month 0, 2, and 4. If 7-23 months of age, vaccination at month 0 and 2. If 2-9 years of age, vaccination at month 0. If patient is HIV positive, vacciation months 0 and 2 if age is 2-9 years.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of 7 - valent pneumococcal conjugated vaccine in HIV - infected children, and assess the predictive factors for protective antibody responses after receiving the vaccine.

DETAILED DESCRIPTION:
S. pneumoniae is an important cause of severe invasive bacterial disease in human immunodeficiency disease (HIV) infected children. The incidence of pneumococcal bacteremia cases requiring hospitalization among Thai children aged < 5 years had a range of 10.6-28.9 cases per 100,000 persons.[1]

Children infected with HIV have a markedly increased risk for pneumococcal infection compared with those who are not HIV-infected. HIV-infected children had rates of invasive pneumococcal disease (IPD) that were 2.8 and 12.6 times the rate among HIV-negative children aged <5 and <3 years, respectively. Incidence of IPD is 6.1 cases/100 patient-years among HIV-infected children through age 7 years [2]

Recent important strategy in prevention of invasive pneumococcal disease (IPD) is an implementation of pneumococcal conjugate vaccine (PCV), which can induce immunity starting from 2 months of age. In a small study of 5-valent PCV among children < 2 years of age, serotype-specific IgG antibodies (ELISA) response after 3 doses was found to be immunogenic among both groups.[3] The Pediatric AIDS Clinical Trials Group Study 292 show that the immunologic responses to 7- valent PCV were similar for all serotypes among asymptomatic and symptomatic HIV - infected children.[4] The study of quantitative and qualitative antibody responses to 9 - valent PCV in HIV-infected children in South Africa shows similar quantitative antibody responses but poorer qualitative antibody responses to the pneumococcal conjugate vaccine when compared to HIV-negative children.[5].

In Thailand, 7 - valent PCV (Prevnar® ) was available in 2003. It is recommended for young children and highly recommended for high risk children such as HIV-infected children, congenital heart disease or premature infants. However, one of the major obstacles for large scale implementation is cost issue. There is no previous study about immunogenicity, safety or efficacy of 7 - valent PCV in HIV -infected Thai children, the objective of this study is to assess the safety and immunogenicity of a 7 - valent PCV vaccine among HIV - infected compared with HIV - exposed children.

ELIGIBILITY:
Inclusion Criteria:

1. HIV - infected children

   * HIV infected individuals
   * Age between 2 months to 9 years
   * Signed written informed consent
2. HIV - exposed negative children

   * Maternal HIV infection, documented prior to delivery.
   * Age between 2 months to 9 years
   * Signed written informed consent

Exclusion Criteria:

* Active opportunistic infection
* History of hypersensitivity to pneumococcal conjugate vaccine or diphtheria toxoid
* Using oral steroid or immunosuppressive drugs
* Received pneumococcal conjugate vaccine, or pnuemococal polysaccharide vaccine

Ages: 2 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
immunogenicity | 28 days
  Proportion of children with PCV serotype - specific IgG antibody at 28 days after completion of primary series of vaccination.

SECONDARY OUTCOMES:
Safety | 28 days
  Number of adverse events after PCV administration
compare serotype | 28 days
  Compare proportion of PCV serotype - specific IgG antibody in HIV - infected children by baseline clinical staging, CD4 and viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Chitsanu Pancharoen, MD, Principal Investigator — Pediatric infectious diseases unit, Chulalongkorn University
Locations (2):
- Thailand (2):
  - HIV-NAT, The Thai Red Cross AIDS Research Center, Bangkok
  - Pediatric infectious diseases section, King Chulalongkorn Memorial hospital, Bangkok

REFERENCES:
- [Result] Thanee C, Pancharoen C, Likitnukul S, Luangwedchakarn V, Umrod P, Phasomsap C, Apornpong T, Chuanchareon T, Butterworth O, Puthanakit T. The immunogenicity and safety of pneumococcal conjugate vaccine in human immunodeficiency virus-infected Thai children. Vaccine. 2011 Aug 11;29(35):5886-91. doi: 10.1016/j.vaccine.2011.06.072. Epub 2011 Jul 3. PMID 21729732
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org